CLINICAL TRIAL: NCT03998631
Title: Comparison of Carbon Dioxide Flush and Saline Flush to Saline Flush Alone in TEVAR and TAVI Procedures to Reduce Cerebral Ischemia
Brief Title: Comparison of Carbon Dioxide and Saline Flush to Saline Flush in TEVAR and TAVI Procedures to Reduce Cerebral Ischemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kongteng Tan, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-5219
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Thoracic Aortic Aneurysm; Aortic Stenosis Symptomatic; Stroke, Complication
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Stroke | interventions — Carbon Dioxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Saline Flush (Placebo Comparator): This is the control arm. The TEVAR or TAVI device will be flushed with at least 60mL of standard saline to reduce bubbles in the reservoir prior to deployment. This is the standard of care.
  Interventions: Procedure: Standard Saline Flush
- Carbon Dioxide and Saline Flush (Experimental): Carbon dioxide flush of the TEVAR or TAVI device followed by saline flush.
  Interventions: Procedure: Carbon Dioxide and Saline Flush

INTERVENTIONS:
Procedure: Carbon Dioxide and Saline Flush — The TEVAR or TAVI device will be flushed with approximately 1.2L of medical grade carbon dioxide using a 60mL syringe and connecting tubing. The reservoir will then be flushed with at least 60mL of standard saline prior to deployment to minimize bubbles in the saline.
  Other Names: Cook Zenith alpha thoracic endovascular graft; Sapien Transcatheter Heart Valve; CoreValve Trascatheter Aortic Valve
  Arms: Carbon Dioxide and Saline Flush
Procedure: Standard Saline Flush — Standard of care flushing of the TEVAR or TAVI device with normal saline.
  Other Names: Cook Zenith alpha thoracic endovascular graft; Sapien Transcatheter heart valve; Core Valve Transcatheter Aortic Valve
  Arms: Saline Flush

SUMMARY:
Thoracic endovascular repair (TEVAR) and transcatheter aortic valve implantation (TAVI) are standard of care procedures to treat thoracic aortic aneurysm or severe aortic stenosis, respectively. Both procedures have a high risk of stroke and silent infarction. Gas has been detected in the cerebral vasculature during these procedures and associated with DWI positive lesions on MRI. The hypothesis is that air emboli contribute to stroke and silent infarction. The investigators propose addressing air emboli by flushing the device with carbon dioxide prior to flushing with saline. This is a pilot study comparing standard saline flush alone to carbon dioxide flushing with saline flush.

ELIGIBILITY:
Inclusion Criteria:

* Elective TEVAR or TAVI
* Over 18 years old

Exclusion Criteria:

* Recent acute myocardial infarction
* Recent stroke or TIA
* Post or pending organ transplantation
* Active peptic ulcer disease
* Recent gastrointestinal bleed
* History of bleeding diathesis or coagulopathy or contraindications to antiplatelet or anticoagulant therapy.
* Permanent pacemaker or ICD
* History of atrial fibrillation
* Moderate or severe allergy to iodinated contrast not amenable to predmedication
* Renal failure
* Unable to safely undergo MRI
* Enrollment in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Complications | 30 days
  Infection, bleeding, stroke, pseudoaneurysm formation, etc.
All cause mortality | 30 days
  Post procedural death.

SECONDARY OUTCOMES:
Stroke | 7 days
  Physical examination and magnetic resonance imaging (MRI) brain.
Silent Infarction | 7 days
  MRI brain.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers.

REFERENCES:
- [Background] Gutsche JT, Cheung AT, McGarvey ML, Moser WG, Szeto W, Carpenter JP, Fairman RM, Pochettino A, Bavaria JE. Risk factors for perioperative stroke after thoracic endovascular aortic repair. Ann Thorac Surg. 2007 Oct;84(4):1195-200; discussion 1200. doi: 10.1016/j.athoracsur.2007.04.128. PMID 17888969
- [Background] Bechara CF. Commentary: Eliminating Air From Stent-Grafts During Arch Endovascular Therapy: One Step Closer to Reducing Stroke. J Endovasc Ther. 2019 Feb;26(1):81-82. doi: 10.1177/1526602818819922. Epub 2018 Dec 21. No abstract available. PMID 30572774
- [Background] Lansky AJ, Brown D, Pena C, Pietras CG, Parise H, Ng VG, Meller S, Abrams KJ, Cleman M, Margolis P, Petrossian G, Brickman AM, Voros S, Moses J, Forrest JK. Neurologic Complications of Unprotected Transcatheter Aortic Valve Implantation (from the Neuro-TAVI Trial). Am J Cardiol. 2016 Nov 15;118(10):1519-1526. doi: 10.1016/j.amjcard.2016.08.013. Epub 2016 Aug 23. PMID 27645761
- [Background] Perera AH, Rudarakanchana N, Monzon L, Bicknell CD, Modarai B, Kirmi O, Athanasiou T, Hamady M, Gibbs RG. Cerebral embolization, silent cerebral infarction and neurocognitive decline after thoracic endovascular aortic repair. Br J Surg. 2018 Mar;105(4):366-378. doi: 10.1002/bjs.10718. Epub 2018 Feb 12. PMID 29431856
- [Background] Rohlffs F, Tsilimparis N, Saleptsis V, Diener H, Debus ES, Kolbel T. Air Embolism During TEVAR: Carbon Dioxide Flushing Decreases the Amount of Gas Released from Thoracic Stent-Grafts During Deployment. J Endovasc Ther. 2017 Feb;24(1):84-88. doi: 10.1177/1526602816675621. Epub 2016 Oct 26. PMID 27798380
- [Background] Kolbel T, Rohlffs F, Wipper S, Carpenter SW, Debus ES, Tsilimparis N. Carbon Dioxide Flushing Technique to Prevent Cerebral Arterial Air Embolism and Stroke During TEVAR. J Endovasc Ther. 2016 Apr;23(2):393-5. doi: 10.1177/1526602816633705. Epub 2016 Feb 19. PMID 26896417
- [Result] Cheng D, Martin J, Shennib H, Dunning J, Muneretto C, Schueler S, Von Segesser L, Sergeant P, Turina M. Endovascular aortic repair versus open surgical repair for descending thoracic aortic disease a systematic review and meta-analysis of comparative studies. J Am Coll Cardiol. 2010 Mar 9;55(10):986-1001. doi: 10.1016/j.jacc.2009.11.047. PMID 20137879